CLINICAL TRIAL: NCT04871282
Title: RINGSIDE: A Phase 2/3, Randomized, Multicenter Study to Evaluate AL102 in Patients With Progressing Desmoid Tumors
Brief Title: A Study of AL102 in Patients With Progressing Desmoid Tumors
Acronym: RINGSIDE
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Immunome, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AL-DES-01
Record Dates: First submitted 2021-04-23; First posted 2021-05-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Desmoid; Desmoid Tumor
Keywords: RINGSIDE
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A Main Study 1.2 mg daily (Experimental): AL102 1.2 mg
  Interventions: Drug: AL102
- Part A Main Study 2 mg Intermittent (Experimental): AL102 2 mg
  Interventions: Drug: AL102
- Part A Main Study 4 mg Intermittent (Experimental): AL102 4 mg
  Interventions: Drug: AL102
- Part B AL102 (Experimental): AL102, recommended dose regimen from Part A, 1.2 mg daily
  Interventions: Drug: AL102
- Part B Placebo (Placebo Comparator): Placebo to match recommended dose regimen from Part A
  Interventions: Other: Placebo
- Open Label Extension (Experimental): AL102, recommended dose regimen from Part A, 1.2 mg daily
  Interventions: Drug: AL102

INTERVENTIONS:
Drug: AL102 — AL102 is an inhibitor of gamma secretase-mediated Notch signaling.
  Other Names: varegacestat
  Arms: Open Label Extension; Part A Main Study 1.2 mg daily; Part A Main Study 2 mg Intermittent; Part A Main Study 4 mg Intermittent; Part B AL102
Other: Placebo — Placebo to match AL102
  Arms: Part B Placebo

SUMMARY:
The current study is designed to evaluate the efficacy and safety of AL102 in patients with progressive desmoid tumors.

DETAILED DESCRIPTION:
This is a Phase 2/3, randomized study in subjects with progressive desmoid tumors consisting of 2 parts. Phase2/Part A is an open-label, dose regimen finding study; Phase3/Part B is a double blind, placebo-controlled study and Open Label Extension utilizing the dose regimen selected in Phase2/Part A.

ELIGIBILITY:
Inclusion Criteria Part A:

1. At least 18 years of age (inclusive) at the time of signing the informed consent form (ICF).
2. Histologically confirmed desmoid tumor (aggressive fibromatosis) by local pathologist (prior to informed consent).
3. Disease progression, assessed locally by the investigator, defined as having at least one of the following:

   * Unidimensional growth of desmoid tumor(s) by ≥10%, using the sum of the largest diameters of target lesion(s), within 18 months of the screening MRI
   * Having desmoid tumor-related pain that is not adequately controlled with nonopioid medication
4. At least 1 measurable lesion amenable to volume measurements by MRI at screening (Part A only)
5. One of the following:

   * Treatment naïve subjects for whom, in the opinion of the investigator, the IP is deemed appropriate, OR
   * Recurrent/refractory disease following at least one line of therapy (including surgery, radiation, or systemic therapy)
6. Agrees to provide formalin-fixed paraffin embedded archival or fresh tumor tissue for re- confirmation of disease.
7. Must be able to swallow whole capsules with no GI condition affecting absorption; nasogastric or G-tube administration is not allowed.

Exclusion Criteria Part A:

1. Diagnosed with a malignancy in the past 2 years with some exceptions.
2. Current or recent (within 2 months of IP administration) GI disease or disorders that increase the risk of diarrhea, such as inflammatory bowel disease and Crohn's disease.
3. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti- fungal therapy ≤7 days prior to administration of IP such as known active infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at Screening.
4. Myocardial infarction within 6 months prior to enrollment, greater than Class 1 angina pectoris, or has New York Heart Association (NYHA) Class III or IV heart failure, , symptomatic ventricular arrhythmias, sustained ventricular tachycardia, Torsade's de Pointes (TdP), the long QT syndrome, pacemaker dependence, or electrocardiographic evidence of acute ischemia.
5. Unstable or severe uncontrolled medical condition (e.g., unstable cardiac or pulmonary function or uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the risk to the subject associated with his or her participation in the study.
6. Pregnant or breastfeeding or expecting to conceive children within the projected duration of the study.
7. Eastern Cooperative Oncology Group (ECOG) performance status ≥2
8. Abnormal organ and marrow function at Screening defined as:

   1. Neutrophils <1000/mm3,
   2. Platelet count <100,000/mm3,
   3. Hemoglobin <9 g/dL,
   4. Total bilirubin >1.5x upper limit of normal (ULN) (except known Gilbert's syndrome),
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >2.5x ULN,
   6. Serum creatinine > ULN and creatinine clearance (CrCl) <60 mL/min (calculation of CrCl will be based on acceptable institution standard)
   7. Uncontrolled triglyceride ≥Grade 2 elevations per common terminology criteria for adverse events (CTCAE) v5.0 (>300 mg/dL or >3.42 mmol/L).
9. ECG Exclusions (Part A only)

   1. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥450 msec.
   2. QRS duration > 110 ms
   3. PR interval > 240 ms
   4. Marked ST-T wave abnormalities which would make it difficult to measure the QT interval
10. Any treatments for desmoid tumors within 4 weeks prior to first dose of investigational therapy; subject must have recovered from therapy related toxicity to < CTCAE Grade 2 or clinical baseline. Therapy includes:

    1. Locoregional tumor directed therapies such as major surgery, radiation, radiofrequency ablation, or cryosurgery
    2. Systemic therapy including chemotherapy, biologic (anti-neoplastic agent, antibodies), TKIs (e.g., sorafenib, pazopanib, imatinib), hormonal therapy, or investigational therapy
11. Chronic NSAIDs for the treatment of desmoid tumors within 4 weeks of first dose of IP;

Inclusion Criteria Part B

1. ≥12 years of age (inclusive) and ≥ 40 kg at the time of signing the ICF.
2. Histologically confirmed desmoid tumor (aggressive fibromatosis) by local pathologist (prior to informed consent) that has progressed by ≥ 20% as measured by RECIST v1.1 within 12 months of the screening visit scan.
3. Evidence of measurable disease by CT/MRI scan. Measurable lesions are defined according to RECIST v1.1.
4. Subject and/or legally authorized representative (i.e. parent/guardian) must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF.
5. Minor subjects must be capable of giving written assent as appropriate per the applicable age (per local regulatory requirements).

For all other inclusion criteria refer to Part A inclusion criteria.

Exclusion Criteria Part B The subjects must be excluded from participating in the study if they meet any of the exclusion criteria for Part A, except where otherwise noted.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Approximately 2 years
  Progression free survival (PFS) as defined as the time from randomization until the date of assessment of progression (as assessed by BICR based on RECIST v1.1) or death by any cause

SECONDARY OUTCOMES:
Overall response rate | Approximately 2 years
  Confirmed overall response rate (ORR) defined as the proportion of subjects with ORR (CR and PR) by BICR based on RECIST v1.1.
Change in Tumor Volume | Approximately 2 years
  Change from baseline in estimated tumor volume measured by T2 weighted (T2W) MRI or CT by BICR (based on RECIST v1.1)
Duration of response | Approximately 2 years
  Duration of response defined by the time from confirmed CR or PR (by BICR based on RECIST v1.1) until the earlier of the first documentation of disease progression or death from any cause.
Progression Free Survival | Approximately 2 years
  Progression free survival (PFS) as defined as the time from randomization until the date of assessment of progression as assessed by BICR (based on RECIST v1.1) or clinical progression as assessed by the investigator or death by any cause
Patient reported outcome | Approximately 2 years
  Change from baseline in pain assessment using GOunder/Desmoid Tumor Research Foundation (DTRF) DEsmoid Symptom Scale and Impact Scale (GODDESS) Desmoid Tumor Symptom Scale (DTSS)
Safety and Tolerability | Approximately 2 years
  Evaluation of the safety and tolerability of AL102 in subjects with progressing desmoid tumors as defined by the frequency and severity of TEAEs and SAEs and the time to treatment discontinuation due to TEAE

CONTACTS AND LOCATIONS:
Overall Officials: Mrinal Gounder, MD, Principal Investigator — MSKCC
Locations (53):
- United States (23):
  - Mayo Clinic, Pheonix, Arizona
  - City of Hope, Duarte, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of California at Los Angeles Hematology/Oncology, Santa Monica, California
  - Stanford University Medical Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - NorthShore University Health System, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Jefferson City Medical Group, Jefferson City, Missouri
  - Washington University, St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UTSW Simmons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Belgium (2):
  - Universitair Ziekenhuis, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
- Germany (2):
  - Helios Klinikum Berlin-Buch, Berlin
  - Mannheim university medical center, Mannheim
- Israel (4):
  - Oncology Institute Barzilai Medical Center, Ashkelon
  - Rambam MC, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (3):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - IRCCS Fondazione Istituto Nazionale dei Tumori, Milan
  - Campus Bio-Medico University Hospital, Rome
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Medisch Centrum, Rotterdam
- Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - ASAN Medical Center, Seoul
- Spain (5):
  - Vall d´Hebrón University Hospital, Barcelona
  - Catalan Institute of Oncology (ICO), Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (4):
  - Western General Hospital, Edinburgh, Scotland
  - Addenbrooke's Hospital, Cambridge
  - The Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No